CLINICAL TRIAL: NCT04181073
Title: The BRAVE Study: Borg Score Outcomes in Respiratory Compromised Acute Exacerbating COPD Patients Receiving Treatment Via Vibrating Mesh Nebuliser Versus Jet Nebuliser in the Emergency Department
Brief Title: Borg Score Outcomes in Respiratory Compromised Acute Exacerbating Chronic Obstructive Pulmonary Disease (COPD) Patients Receiving Treatment Via Vibrating Mesh Nebuliser Versus Jet Nebuliser in the Emergency Department
Acronym: BRAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Clyde and Glasgow (Other)
Collaborators: Aerogen (Industry)
Responsible Party: Principal Investigator, David Lowe, Consultant Emergency Medicine, NHS Greater Clyde and Glasgow
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GN17RM666
Record Dates: First submitted 2019-11-23; First posted 2019-11-29 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: COPD Exacerbation; COPD
Keywords: nebulisation; vibrating mesh nebuliser
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Jet Nebuliser (Active Comparator): Standard therapy of one dose of 0.5 MG Ipratropium and 3 doses of 2.5 MG Salbutamol via Jet Nebuliser
  Interventions: Device: Jet Nebuliser
- Vibrating Mesh Nebuliser (Experimental): Standard therapy of one dose of 0.5 MG Ipratropium and 3 doses of 2.5 MG Salbutamol via Vibrating Mesh Nebuliser
  Interventions: Device: Vibrating Mesh Nebuliser

INTERVENTIONS:
Device: Jet Nebuliser — Jet Nebuliser
  Arms: Jet Nebuliser
Device: Vibrating Mesh Nebuliser — Aerogen Device
  Arms: Vibrating Mesh Nebuliser

SUMMARY:
The purpose of this study is to compare clinical outcomes in patients with acute COPD treated with a vibrating mesh nebuliser (VMN) versus a current standard jet nebuliser (JN), in the Emergency Department (ED).

Participants will be those who meet the inclusion criteria and have a primary diagnosis of COPD, and consent to take part in the study. Operators will be clinical staff including doctors and nurses who will be trained in the use of the nebulisers.

Delivery of current treatment standards utilising a VMN compared to a JN will improve symptom scores in patients attending ED with COPD exacerbations.

DETAILED DESCRIPTION:
This study is a prospective, single-centre, open, randomised study to improve management of acute COPD exacerbation within the Emergency Department. Adults with severe COPD are randomised into 2 groups: vibrating mesh nebuliser or standard jet nebuliser treatment. Salbutamol (5mg) and Ipratropium (0.5mg) will be administered via Aerogen Ultra via valved mask or a standard jet nebuliser via open face mask/. Two further doses of salbutamol to be delivered.

ELIGIBILITY:
Inclusion Criteria:

* • Primary presentation with acute exacerbation of COPD

Exclusion Criteria:

* • Unable to give valid consent

  * Patient unable to speak English
  * Patients where alternative diagnosis cannot be excluded
  * Known or suspected pneumonia, pneumothorax, pneumomediastinum, pulmonary oedema, vocal cord dysfunction, aspirated foreign body
  * Any contraindication to delivering bronchodilators
  * Need for immediate intubation , ventilation or non-invasive ventilation
  * Pregnant or lactating
  * Active palliation considered or expected mortality within 48 hours
  * Known background/ comorbid respiratory disease associated with chronic or variable airflow obstruction (significant goitre, central lung tumour or other central airway pathology, bronchiectasis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
BORG Score | 30 minutes post treatment
  Change in Reported Dyspnoea. Modified BORG dyspnoea scale. 0 (best) min 10 max (worse)

SECONDARY OUTCOMES:
Oscillometry | 30 minutes post treatment
  Change of Oscillometry data
Escalation of Care | During Emergency Department Admission (typically < 4 hours)
  Requirement for NIV (non invasive ventilation) / Intubation / further nebulisation
Blood Gas | 30 minutes post treatment
  Change in blood gases post treatment
Completion of Treatment | During Emergency Department Admission (typically < 4 hours)
  Time to complete initial nebulisation therapy in ED
Staff Satisfaction | During Emergency Department Admission (typically < 4 hours)
  Reported ED staff satisfaction from main care giver post treatment. Likert 5 point scale. (0 highly dissatisfied 5 highly satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored in Safe Haven GG&C
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: Via Safe Haven Committee